CLINICAL TRIAL: NCT03476512
Title: Treatment Adherence and Blood Pressure Outcome Among Hypertensive Out-patients in Two Tertiary Hospitals in Sokoto, Northwestern Nigeria
Brief Title: Treatment Adherence and Blood Pressure Outcome Among Hypertensive Out-patients
Status: Completed | Type: Observational
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, DR RASAQ ADISA, Director, Medication Therapy Management Research in Communicable and non-communicable, University of Ibadan
Other Study IDs: TAHYP001
Record Dates: First submitted 2018-02-28; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: Treatment adherence; Ambulatory hypertensive patients; Blood pressure; Non-pharmacological measures
MeSH Terms: conditions — Hypertension; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adherence Education — Patients were given adherence education to resolve the identified deficits

SUMMARY:
It is estimated that more than 70% of patients on antihypertensive medications do not take them as prescribed. Treatment non-adherence practice may be particularly higher in developing countries where there is poor accessibility to medicines and healthcare services, coupled with low level of awareness of the lifelong nature of hypertension treatment among patients. Optimal control of blood pressure has been reported to reduce the incidence of morbidity and mortality associated with hypertension. Thus, adoption of healthy lifestyle as well as ensuring regular and continuous adherence to prescribed medications are integral to successful management of hypertension to achieve the target blood pressure goals.

The present study comprehensively evaluated adherence to pharmacotherapy and non-pharmacological measures among ambulatory hypertensive patients attending two healthcare institutions in Sokoto, Northwestern Nigeria. Reasons for treatment non-adherence were evaluated, while perception and beliefs about hypertension and its management were also explored, with pharmacist-led patient-specific adherence education provided as appropriate to resolve the knowledge gap(s). Association between treatment adherence and blood pressure outcome at contact and the subsequent 2-months clinic appointment were investigated.

Patients aged 18 years and above, with a primary diagnosis of hypertension, and who were on antihypertensive medications for at least 3-months were recruited from the medical outpatient clinic of Usmanu Danfodiyo University Teaching Hospital and the Specialist Hospital, both within Sokoto metropolis, Sokoto state, Northwestern Nigeria. Newly diagnosed patients, in-patients and those who declined participation were excluded from the study.

DETAILED DESCRIPTION:
Background: Hypertension is a common cardiovascular disease worldwide, contributing 4.5% of the global disease burden and 12.8% premature deaths annually. Despite recent advances in drug therapy, majority of diagnosed hypertensive patients are poorly controlled. Reasons for inadequate control of hypertension are heterogeneous including low adherence to antihypertensive medications and lifestyle changes, low compliance with scheduled follow-up visits and suboptimal pharmacotherapy. This study evaluated adherence to pharmacotherapy and non-pharmacological measures among ambulatory hypertensive patients, reasons for treatment non-adherence were evaluated, while perception and beliefs about hypertension and its management were also explored, with pharmacist-led patient-specific adherence education provided as appropriate to resolve the knowledge gap(s). Association between treatment adherence and blood pressure outcome at contact and the subsequent 2-months clinic appointment were investigated.

Method: This study involved a cross-sectional questionnaire-guided interview and retrospective review of medical records of 605-patients from two hospitals. Nine-item modified adherence predictor scale was used to assess medication adherence. Overall adherence score to lifestyle modifications was obtained from the total scores from 4-domains of non-pharmacological measures including cigarette smoking and alcohol cessation, salt-restriction and exercise. Patient-specific adherence education was provided at contact to resolve the knowledge gap(s). Clinical-parameters especially the blood pressure values were retrieved at contact and subsequent 2-months appointment. Data were summarised using frequency, percentage, 50th percentile and mean ± standard deviation. Chi-square test was used to evaluate association between socio-demographic variables and adherence to antihypertensive medication and lifestyle recommendations. Student's t-test was used to investigate relationship between treatment adherence and blood pressure outcome at p < 0.05 considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above, with a primary diagnosis of hypertension, and who were on antihypertensive medications for at least 3-months were enrolled.

Exclusion Criteria:

* Newly diagnosed patients, in-patients and those who declined participation were excluded from the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory hypertensive patients
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Questionnaire with a nine-item adherence scale to assess the level of adherence to medication | 5 hours on Thursday clinic days, 16 weeks
  Questionnaire with a nine-item adherence scale was used to assess the level of adherence to medication, while dichotomous Yes/No response option was used to evaluate the level of adherence to the 4-domains of non-pharmacological lifestyle modifications, specifically smoking, alcohol, exercise, and salt-restriction. Using the Statistical Package for Social Sciences version 22 at p < 0.05 level of significance, descriptive statistics including frequency and percentage was used to summarise the data on these parameters

SECONDARY OUTCOMES:
Perception and belief about hypertension and treatment | 5 hours on Thursday clinic days, 16 weeks
  Modified Brief Illness Perception Questionnaire, and 9-item Belief bout Medicine Questionnaire with a 5-point likert scale was used to evaluate the perception and belief of patients about hypertension and the treatment. Descriptive statistics including frequency, percentage and 50th percentile was used to summarise the data on perception and belief about hypertension and treatment, using the Statistical Package for Social Sciences version 22.
Data collection form to retrieve the average of two consecutive blood pressure readings (Systolic and Diastolic) | 4 hours on Thursday clinic days, 16 weeks
  Data collection form was designed to retrieve the average of two consecutive blood pressure readings (Systolic and Diastolic) in individual patient's case note at contact and at the 2-months clinic appointment. Descriptive statistics including frequency, mean ± standard deviation was used to summarise these continuous variable data Chi-square and student's t-test were used to evaluate the relationship between treatment adherence and blood pressure outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Usmanu Danfodiyo University Teaching Hospital, Sokoto, Nigeria